CLINICAL TRIAL: NCT04231279
Title: A Phase II Study to Identify the Role of Exocrine Pancreatic Insufficiency in Pediatric Patients With Abdominal Pain (RAP) Who Are Undergoing Upper Endoscopy Using Synthetic Human Secretin
Brief Title: Recurrent Abdominal Pain and Exocrine Pancreatic Insufficiency
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data collection discontinuity and sponsor reallocation of study resources to manufacturing
Sponsor: Orlando Health, Inc. (Other)
Collaborators: ChiRhoClin, Inc. (Industry)
Responsible Party: Principal Investigator, Devendra Mehta, Director, Pediatric Gastroenterology Laboratory, Arnold Palmer Hospital for Children, Orlando Health, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RAP and EPI; 1804804 (Other: Orlando Health IRB #2)
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Pain; Irritable Bowel Syndrome
MeSH Terms: conditions — Abdominal Pain; Irritable Bowel Syndrome | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ChiRhoStim Group 1 (Active Comparator): Patients undergoing EGD with ePFT for symptoms of suspected or known pancreatic insufficiency.
  Interventions: Drug: synthetic human secretin
- ChiRhoStim Group 2 (Experimental): Patients undergoing diagnostic EGD that consent to undergo ePFT.
  Interventions: Drug: synthetic human secretin

INTERVENTIONS:
Drug: synthetic human secretin — Secretin is a gastrointestinal peptide hormone, indicated for the stimulation of: pancreatic secretions, including bicarbonate, to aid in the diagnosis of pancreatic exocrine dysfunction.
  Other Names: ChiRhoStim

SUMMARY:
This is a 3-year prospective study too identify the role of exocrine pancreatic insufficiency in patients with abdominal pain who are undergoing upper endoscopy. An endoscopic pancreatic function test (ePFT) with secretin will be performed in children undergoing routine investigative EGD.

The goal of this study is to identify the role of exocrine pancreatic insufficiency in patients with abdominal pain who are undergoing upper endoscopy, who otherwise would be labelled as recurrent abdominal pain (RAP).

DETAILED DESCRIPTION:
Recurrent abdominal pain (RAP) is an often encountered complaint in children and adolescents. The evaluation of the child or adolescent with recurrent abdominal pain requires an understanding of the pathogenesis of abdominal pain, the most common causes of abdominal pain, and the typical patterns of presentation.

Children and adolescents frequently undergo esophagogastroduodenoscopy (EGD) to evaluate complaint and recurrent abdominal pain is a frequently cited reason for endoscopy. This is a standard procedure where an endoscope is passed through the mouth, esophagus, stomach and into the first part of the small intestine. With the camera at the end of the endoscope, the endoscopist is able to see the gross appearance of the upper digestive tract. Small biopsy samples are collected from the small intestine, stomach and esophagus to evaluate for mucosal injury, irritation, infection or other anomalies that could be contributing to the patient's symptoms. This is helpful for evaluation of histological changes, but does not provide information about its function.

Pancreatic stimulation testing with secretagogue (secretin, cholecystokinin) administration, and direct pancreatic fluid collection is considered a gold standard to assess the exocrine pancreatic function. Indirect testing of pancreatic function such as with urine or stool has much lower sensitivity and specificity compared to direct pancreatic fluid collection.

This is a prospective study where patients undergoing investigative EGD will have endoscopic pancreatic function test (ePFT) with secretin.

There will be two groups:

The first group are patients that are undergoing EGD with ePFT for evaluation of suspected or established pancreatic insufficiency with symptoms such as failure to thrive or malabsorption. These patients are the ones that historically have had ePFT testing done to evaluate their pancreatic function.

The second group is all patients that are undergoing scheduled diagnostic EGD for other reasons that consent for pancreatic stimulation testing. These patients are usually undergoing EGD for a range of symptoms that frequently include recurrent abdominal pain, bloating, diarrhea, nausea and/or constipation. These patients do not typically have ePFT testing performed and is not usually thought to be part of the standard of care for this group.

ELIGIBILITY:
Inclusion Criteria:

* For Group 1- Patients undergoing EGD with ePFT for symptoms of suspected or known pancreatic insufficiency
* For Group 2- Patients undergoing diagnostic EGD who consent to undergo ePFT

Exclusion Criteria:

* If it is an emergency EGD procedure
* If the caregiver refuses to sign the consent form
* Patient has undergone ePFT testing previously with a documented allergy to human secretin
* Patients that require atropine at the time of sedation

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of pancreatic insufficiency in Pediatric cases undergoing upper endoscopy for Abdominal Pain | 2.5 years
  Secretin stimulated exocrine pancreatic enzyme activity will be measured in patients with abdominal pain who are undergoing upper endoscopy to identify those with insufficiency (EPI).

SECONDARY OUTCOMES:
Secondary biomarkers for exocrine pancreatic insufficiency in blood and pancreatic fluid will be measured to explore mechanisms involved leading to abdominal pain and become potential tests in future. | 2.5 years
  This includes immunological and genetic markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health - Arnold Palmer Children's Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No